CLINICAL TRIAL: NCT04645173
Title: A Multi-Center Study Evaluating Participants Who Received CanGaroo® Envelope, TYRX™ Envelope, or No Envelope During CIED Implantation
Brief Title: Comparison of Participants Who Received a CanGaroo® Envelope, TYRX™ Envelope, or no Envelope During CIED Implantation
Acronym: HEAL
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR-2214
Record Dates: First submitted 2020-11-16; First posted 2020-11-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Characteristics of soft tissue healing surrounding the CIED implant as assessed by blinded histologic evaluation of systematic biopsies taken at the time of change-out/revision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- CanGaroo Envelope: Participants who received a CanGaroo envelope during CIED implantation
  Interventions: Device: CIED envelope
- TYRX Envelope: Participants who received a TYRX envelope during CIED implantation
  Interventions: Device: CIED envelope
- No Envelope: Participants who did not receive an envelope during CIED implantation

INTERVENTIONS:
Device: CIED envelope — Evaluation of the difference in cohorts for soft tissue healing surrounding the CIED implant and clinical outcomes and complications.
  Groups: CanGaroo Envelope; TYRX Envelope

SUMMARY:
The objective of this study is to gather information on participants returning at time of CIED change-out or revision who underwent a device implantation with either a CanGaroo® envelope, TYRX™ envelope, or no envelope.

DETAILED DESCRIPTION:
This multi-center study will enroll up to approximately 100 participants who have undergone one or more implantations of a CIED with either CanGaroo®, TYRX™, or no envelope (up to approximately 30-35 participants per cohort) and are returning for a CIED change-out or revision procedure at least 4 months or longer from their prior procedure.

Once enrolled, each participant will have their medical history data collected (baseline demographics, medical history, prior CIED exchanges/revisions, and post implant clinical events). Prior to the scheduled change-out/revision procedure, there will be an assessment of the current healed implant site skin incision independently by both the participant and investigator using the Patient and Observer Scar Assessment Scale (POSAS), as well as photographs taken of the current skin scar.

During the change-out/revision procedure, additional investigator assessments will include photographic documentation of CIED implant pocket lining, classification of the extent of lead adhesions in the implant pocket, and biopsies of the anterior and posterior capsule walls for histologic analysis. Procedural details and any complications/AEs that occur during the change-out/revision procedure will also be captured.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who previously underwent one or more prior CIED implantations utilizing a CanGaroo® envelope, TYRX™ envelope, or no envelope and are returning for a CIED change-out or revision procedure at least 4 months or longer from their prior procedure.
2. The following possible scenarios would be eligible for enrollment:

   a. One prior CIED Implant: i. No envelope ii. CanGaroo® envelope iii. TYRX™ envelope b. Multiple prior CIED Implants (envelope type should remain the same for each participant throughout their implant history): i. No envelope → no envelope ii. No envelope → CanGaroo® envelope iii. No envelope → TYRX™ envelope iv. CanGaroo® envelope → CanGaroo® envelope v. TYRX™ envelope → TYRX™ envelope vi. No envelope → CanGaroo® envelope → CanGaroo® envelope vii. No envelope → no envelope → CanGaroo® envelope viii. No envelope → TYRX™ envelope → TYRX™ envelope ix. No envelope → no envelope → TYRX™ envelope
3. Participants aged 18 years or older at time of enrollment.
4. Participant is able and agrees to provide written informed consent and use of PHI.
5. Participants for whom prior CIED implant history information can be obtained.

Exclusion Criteria:

1. Active infection involving the CIED implant site (clinical diagnosis of an active infection at the time of change-out/revision procedure).
2. Participants under the age of 18 at time of enrollment.
3. Participants with a history of multiple prior CIED implants over time using more than one type of envelope will be excluded as well as participants with a history of one type of envelope use, but the current pocket does not have an envelope. Scenarios that would be excluded:

   1. CanGaroo® envelope → TYRX™ envelope
   2. TYRX™ envelope → CanGaroo® envelope
   3. CanGaroo® envelope - no envelope
   4. TYRX™ envelope → no envelope
   5. No envelope → CanGaroo® envelope → no envelope
   6. No envelope → TYRX™ envelope → no envelope
   7. No envelope → CanGaroo® envelope → TYRX™ envelope
   8. No envelope → TYRX™ envelope → CanGaroo® envelope
   9. CanGaroo® envelope → no envelope → TYRX™ envelope
   10. TYRX™ envelope → no envelope → CanGaroo® envelope
   11. CanGaroo® envelope → TYRX™ envelope → no envelope
   12. TYRX™ envelope → CanGaroo® envelope → no envelope
   13. CanGaroo® envelope → CanGaroo® envelope → no envelope
   14. TYRX™ envelope → TYRX™ envelope → no envelope
4. Participants undergoing a change-out or revision procedure less than 4 months from their prior procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who underwent one or more prior CIED implantation procedure at the current implant site utilizing CanGaroo®, TYRX™, or no envelope and are returning for a CIED change-out or revision procedure.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Blinded Histologic Evaluation of Biopsies Taken from the Anterior and Posterior Capsule Wall | Surgical Procedure Visit
  Microscopic analysis of cellularity, vascularity, collagen density, necrosis, infectious agents, remnant device material, giant cells, and fibrotic capsule thickness will be evaluated for each biopsy site using a quantitative scoring system with an attempt to distinguish between remnant envelope collagen (if ECM envelope was used) and neocollagen from the participant. Composite (total) and average scores will be determined based on the individual scores from each biopsy site. The quantitative thickness of each fibrotic capsule biopsy will be measured using digital image software. Four (4) thickness measurements will be performed across the image for each biopsy sample, and the average fibrotic thickness will be reported for each sample. In addition, the total average thickness across the four samples will be determined based on the average individual recordings.

SECONDARY OUTCOMES:
Documented CIED Complications | Pre-Surgery Visit
  Comparison between cohorts of documented clinical outcomes and complications since the most recent CIED procedure through the current change-out/revision procedure. Assessment of the clinical outcomes & events of the 3 cohorts will inform on potential differences in clinical outcomes that may be related to the cohort treatment. For example: infection, Twiddler's syndrome, CIED migration, CIED erosion, lead revision, lead dislodgement, pocket revision, device reprogramming, pocket revision.

OTHER OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | Pre-Surgery Visit
  10-point score: Each item of the POSAS is rated on a 10-point score. The lowest score is '1', which corresponds to the situation of normal skin (i.e., normal pigmentation, no itching). Score 10 equals the largest difference from normal skin (i.e., the worst imaginable scar or sensation).
  Total score: The total score of both scales can be simply calculated by summing up the scores of each of the six items. The total score can range from 6 to 60. The overall opinion item is not included in the sum score.
CIED Scar Photographs | Pre-Surgery Visit
  Comparison of photographs of the previous skin incision scar taken pre-surgery. The visual differences in the skin incision scar appearance between the 3 cohorts may correlate with histologic findings and/or post-implant clinical outcomes or events.
CIED Implant Photographs | Surgical Procedure Visit
  Comparison of photographs of the previous CIED implant pocket interior taken intraoperatively. The visual differences in interior capsule wall appearance between the 3 cohorts may correlate with histologic findings and/or post-implant clinical outcomes or events.
Assessment of Lead Adhesions within the Implant Pocket | Surgical Procedure Visit
  * This observation should be made while the CIED device is mobilized and removed from within the implant pocket.
  * The classification system is based on two estimated factors:
    * The amount of fibrosis by visual estimate (none/trivial, mild, moderate, or severe).
  NOTE: If calcification is present, the capsule should be classified as Class 3 (severe).
  * The estimate of the percentage of the lead coiled within the implant pocket that is adhered or trapped within the capsule wall (Class 0: none, Class 1: <30%, Class 2: 30%-60%, and Class 3: >60%).

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Valley Heart Rhythm Specialists, Chandler, Arizona
  - Bay Pines VA, Bay Pines, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida
  - Prairie Education & Research Cooperative / St. John's Hospital, Springfield, Illinois
  - U of L Health/Jewish Hospital, Louisville, Kentucky
  - Columbia University Irving Medical Center, New York, New York
  - Atrium Health, Concord, North Carolina
  - East Carolina University/Vidant Medical Center, Greenville, North Carolina
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aziyo Biologics, Inc. — http://aziyo.com